CLINICAL TRIAL: NCT02144636
Title: Effect of Protein Supplementation on Weight Loss and Cardio Metabolic Profile of Overweight/Obese Subjects
Brief Title: Protein Supplementation and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: herbalife.2014
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treament (Experimental): herbalife protein shake along with exercise
  Interventions: Dietary Supplement: herbalife protein shake
- control (No Intervention): diet and exercise only

INTERVENTIONS:
Dietary Supplement: herbalife protein shake
  Arms: treament

SUMMARY:
This randomized control trial of diet with protein supplementation is being conducted to test the hypothesis that in overweight/obese subjects high protein diet may lead to weight loss and improvement in cardio-metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 21 -65 years
2. Subjects with BMI > 23 Kg/m2

Exclusion Criteria:

* Inclusion Criteria:

  1. Subjects aged between 21 -65 years
  2. Subjects with BMI > 23 Kg/m2

Exclusion Criteria:

1. Diabetes (type 1 and type 2)
2. Known or documented coronary heart disease (CHD) (including ECG consistent with prior myocardial infraction), cerebrovascular accident (including transient ischemic attack), peripheral vascular disease (including symptoms of claudication)
3. Angina or other chest pain that may indicate CHD by history
4. Clinically significant neoplastic, cardiovascular, hepatic, renal, metabolic, endocrine (untreated or unstable), or psychiatric (untreated or unstable) by history
5. Medications: Lipid lowering therapy, daily NSAID or greater than 325 mg ASA (PRN use ok), clopidogrel (or equivalent), Coumadin, other investigational drugs within 30 days of study entry
6. Pregnancy or planning pregnancy during the study period by history
7. Uncontrolled hypertension
8. Uncontrolled hypothyroidism
9. Sensitivity or allergy to product by history
10. Subjects who had undergone bypass procedure
11. Any debilitating disease such as tuberculosis, HIV by history .
12. Unwillingness to give written informed consent for participation in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
weight loss | baseline to 3 months

SECONDARY OUTCOMES:
improvement in lipid profile | baseline - 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fortis-C-DOC Centre of Excellence for Diabetes, Metabolic Diseases and Endocrinology, Delhi, India